CLINICAL TRIAL: NCT01784042
Title: Effect of Dietary Energy Restriction and Omega-3 Fatty Acids on Mammary Tissue and Systemic Biomarkers of Breast Cancer Risk
Brief Title: Dietary Energy Restriction and Omega-3 Fatty Acids on Mammary Tissue
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Manni, Professor and Chief, Division of Endocrinology, Diabetes and Metabolism, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 12-075
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; omega-3 fatty acids
MeSH Terms: conditions — Breast Neoplasms | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No dietary energy restriction plus Placebo (Placebo Comparator): No dietary energy restriction plus Placebo
  Interventions: Drug: Placebo
- Dietary energy restriction plus placebo (Placebo Comparator): Dietary energy restriction plus placebo
  Interventions: Drug: Placebo; Other: Dietary energy restriction
- Lovaza (Experimental): Lovaza only
  Interventions: Drug: Lovaza
- Dietary energy restriction plus Lovaza (Experimental): Dietary energy restriction plus Lovaza
  Interventions: Drug: Lovaza; Other: Dietary energy restriction

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Dietary energy restriction plus placebo; No dietary energy restriction plus Placebo
Drug: Lovaza
  Other Names: Lovaza (omega-3-acid ethyl esters)
  Arms: Dietary energy restriction plus Lovaza; Lovaza
Other: Dietary energy restriction
  Arms: Dietary energy restriction plus Lovaza; Dietary energy restriction plus placebo

SUMMARY:
The over-reaching goal of this study is to test the merit of combining dietary energy restriction with omega-3 fatty acids as a safe and effective breast cancer chemoprevention strategy in overweight and obese women at high risk.

DETAILED DESCRIPTION:
Obesity over the pre- and postmenopausal years is linked to the risk of postmenopausal breast cancer. Multiple mechanisms are likely to contribute to obesity associated breast cancer risk. They include increased insulin like growth factor (IGF)-I bioavailability, oxidative stress, raised leptin to adiponectin ratio, and increased inflammatory cytokines which are responsible for the creation of a systemic and local hyperestrogenic milieu by induction of aromatase and may also be responsible for the reduction in antitumor immunity by stimulation of immunosuppressive cells. While derivative chromosome disulfiram (DER) has been shown to reverse some of these obesity related phenotypic features, it is not yet established whether DER reduces breast cancer risk using validated tissue biomarkers predictive of breast cancer development. N:3FA (3-fatty acids) have been shown to ameliorate obesity-induced effects on circulating leptin and adiponectin, insulin resistance, endogenous estrogen production and inflammation. Although preclinical studies have indicated a protective effect of n:3FA on mammary carcinogenesis, the data in humans are inconclusive, likely as a result of the lack of controlled clinical trials. Investigators hypothesize that the combination of DER and n:3FA will reduce breast cancer risk in an additive/synergistic fashion through their complementary effects on the multiple inter-related pathways accounting for the obesity associated breast cancer risk. Investigators propose to conduct a clinical trial study involving overweight and obese women between the ages of 30 and 55 who are at high risk of breast cancer and are found on random periareolar fine needle aspiration to have hyperplasia with or without atypia with Ki67 ≥2 if premenopausal and ≥1.5 if postmenopausal. Following stratification according to menopausal status they will be randomized to one of four experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Five year predicted breast cancer risk of at least 1.66%.
* Prior breast biopsy showing atypical ductal or lobular hyperplasia or lobular carcinoma in situ or ductal carcinoma in situ (DCIS).
* Known breast cancer-1 and -2 mutations.
* Breast density >50% as assessed by the conventional two-dimensional method.

Exclusion Criteria:

* Weight loss of 10 pounds in past six months.
* History of fish allergy.
* Oral contraceptives or hormone replacement therapy in the past 6 months.
* Pregnancy or lactation in the last 12 months or planning to become pregnant in the next 12 months.
* Current smoking.
* Diagnosis of cancer except basal cell carcinoma of the skin or lobular carcinoma in situ or DCIS.
* Diagnosis of type 1 or type 2 diabetes based on standard criteria, irrespective of treatment.
* Recent stroke or cardiovascular event.
* History of eating disorders documented in medical records.
* History of major gastrointestinal disease impairing absorption.
* History of bariatric surgery.
* Recent, current or planned use of diet drugs as per patient history.
* Participants must not use flaxseed oil supplements during study participation.
* Participants must not use Omega-3 preparations while participating on this trial.
* Participants must not use Tamoxifen or Raloxifene during study participation.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Ki67 expression | about 1 year
  Ki67 expression by hyperplastic breast lesions

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Manni, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States